CLINICAL TRIAL: NCT02677350
Title: A Phase I, Pilot Trial to Evaluate the Safety and Efficacy of Injection of Allogeneic Mesenchymal Bone-Marrow Derived Human Stem Cells in Patients With Fistulizing Crohn's Disease.
Brief Title: AlloGeneic Human Mesenchymal Stem Cells (hMSC) in PAtients With FistuLizing Crohn's Disease Via PErifistula iNjEctions (GALENE)
Acronym: GALENE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study is permanently closed to enrollment
Sponsor: Joshua M Hare (Other)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Sponsor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150965
Record Dates: First submitted 2016-02-01; First posted 2016-02-09 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease; Fistulizing Crohn's Disease; Stem Cells
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pilot (Experimental): Twenty (20) subjects will be treated with 20 million (2 x 10^7) Allogeneic Bone Marrow derived Human Mesenchymal Stem Cells (hMSCs) total divided into 10 injections of 2 million cells/cm of tract in 0.5 ml volume (for total volume of 5 ml per visit) at 4 week intervals for a maximum of 4 treatment sessions based on the discretion of the endoscopist at the time of injection.
  Interventions: Drug: Allogeneic Bone Marrow derived Human Mesenchymal Stem Cells (hMSCs)

INTERVENTIONS:
Drug: Allogeneic Bone Marrow derived Human Mesenchymal Stem Cells (hMSCs) — Peri-fistula injections
  Other Names: allo-hMSCs

SUMMARY:
To evaluate the role of allogeneic mesenchymal stem cells for treatment of perianal fistulizing Crohn disease.

Twenty (20) Crohn's disease patients with complex or multiple perianal or rectovaginal fistulas will be included and will be scheduled to undergo peri-fistula injections after meeting all inclusion/exclusion criteria's at baseline.

Following the Pilot Phase of four (4) subjects, sixteen (16) subjects are scheduled to undergo perianal injections and after meeting all inclusion/exclusion criteria's, will be evaluated at baseline.

DETAILED DESCRIPTION:
Twenty (20) subjects will be treated with 20 million (2 x 10^7) allogeneic MSC's total divided into 10 injections of 2 million cells/cm of tract in 0.5 ml volume (for total volume of 5 ml per visit) at 4 week intervals for a maximum of 4 treatment sessions based on the discretion of the endoscopist at the time of injection..

For patients with more than 6 fistula tracts, the largest of the tracts will be injected.

The first four (4) subjects that receive their initial injections will not be treated less than 5 days apart. As stated in the above response, these first four (4) patients will have an initial safety follow up period of one month prior to proceeding with the treatment of further patients.

Follow up: Clinical (CDAI, PDAI, and perianal examination +/- under anesthesia), and endoscopic ultrasound will be performed at the time of each treatment. MRI evaluation will be performed at screening, 4 weeks after the fourth treatment (week 16) and at 16 months, if fistula closure has not been achieved. Clinical evaluation will be performed at months 1, 3, 6, 12. Endoscopic ultrasound and MRI will also be performed as needed for symptomatic patients if an abscess is suspected.

Duration of Study participation: 17 Months (Follow-up visits will be at 4, 7, 10 and 16 Months post treatment.

The Allo-hMSCs will be supplied from an allogeneic human mesenchymal stem cell source manufactured by the University of Miami.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Male and Female subjects ≥ 18 years of age at the time of signing the Informed Consent Form.
3. Subjects with Fistulizing Crohn´s disease with complex perianal fistula, multiple perianal fistulas, or rectovaginal fistula(s). The complex perianal fistula is defined as a trans-sphincteric, supra-sphincteric or an extra-sphincteric tract. Patients with multiple fistulas, "horseshoe" fistula," or any fistula with fecal incontinence as a result of the Crohn's disease itself or because of previous anal fistula surgery that cannot have more surgery are also eligible.
4. If drainage of abscess is needed, it should be done 2 or more weeks prior to onset of therapy.
5. Have had Crohn's Disease (CD) diagnosed at least 6 months prior to enrollment based on clinical, endoscopic, anatomic/pathologic and/or radiologic criteria.
6. Have a CDAI score <350.
7. During the course of the subject's Crohn's disease (CD), subject must have received anti-Tumor Necrosis Factor (TNF) agents or immunomodulators which did not heal the CD fistulas. If anti-TNFs or immunomodulators are contraindicated or led to adverse events, patients must have failed conservative therapy with antibiotics, or setons, or surgical intervention.
8. Subject who are currently receiving anti-TNFs, antibiotics, 5-aminosalicylic acid, azathioprine, 6-mercaptopurine, methotrexate, prednisone, or any similar drugs at the time of enrollment as long as the following criteria are met:

   1. The patient must have been on the anti-TNF for at least 4 months
   2. The dose of 5-aminosalicylic acid (5-ASA) must have been stable for at least 4 weeks prior to enrollment.
   3. The dose of steroids must have been stable for at least 2 weeks prior to enrollment.
   4. The dose of antibiotics must have been stable for at least 2 weeks prior to enrollment.
   5. The dose of immunomodulators (for example, azathioprine, 6-mercaptopurine, or methotrexate) must have been stable for at least 8 weeks prior to enrollment and the subject on therapy for at least three months prior to enrollment
9. Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements

Exclusion Criteria:

In order to participate in this study, a patient Must Not:

1. Have a known, serious radiographic contrast allergy (gadolinium in particular)
2. Have a hematologic abnormality as evidenced by hematocrit < 25%, white blood cell < 2,500/ul or platelet values < 100,000/ul without another explanation.
3. Have liver dysfunction, as evidenced by enzymes (AST and ALT) greater than three times the Upper limit normal.
4. Have a coagulopathy (International Normalized ratio (INR) > 1.3) not due to a reversible cause (i.e., Coumadin). Patients on Coumadin will be withdrawn 5 days before the procedure and confirmed to have an INR < 1.3. Patients who cannot be withdrawn from Coumadin will be excluded from enrollment.
5. Bone marrow dysfunction, as evidenced by a 20% or more deviation from normal hematocrit, white blood cell count or platelet values without another explanation.
6. Be an organ transplant recipient.
7. Clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
8. Non-cardiac condition that limits lifespan to < 1 year.
9. Patients with a highly active luminal CD, i.e., if they meet any of the following criteria: - Presence of severe proctitis (prominent friability, spontaneous bleeding, multiple erosions, deep ulcers) or very active luminal disease that requires immediate treatment, revealed by colonoscopy.
10. Have anal dysplasia
11. Patients that have received radiation to the pelvic/perianal area.
12. Presence of abscess or other collections not drained (revealed by baseline radiologic study).
13. Presence of setons unless they are removed before treatment beginning.
14. Rectal and/ or anal stenosis that cannot be adequately evaluated for dysplasia by Examination under anesthesia or endoscopy.
15. Need surgery in the perianal region for reasons other than fistulas at inclusion or within 16 weeks after treatment administration.
16. Had a stable dose of an anti-TNF agent within the past 8 weeks before the cell treatment administration.
17. Taking tacrolimus or cyclosporine and not on a stable maintenance dose for 2 weeks before the start of scheduled interventions.
18. Have a history of alcohol or other addictive substances abuse within 6 months before inclusion.
19. Severe uncontrolled diseases (chronic renal failure, cardiovascular, pulmonary or any systemic disease).
20. Any type of medical or psychiatric disease which are considered as exclusion criteria, in the investigator's opinion.
21. Subjects with congenital or acquired immunodeficiency.
22. Positive serology for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV), Human papillomavirus (HPV) or Herpes Virus.
23. Had major surgery or serious traumatism within 6 weeks of enrollment.
24. Impossibility of doing an radiological exploration (reaction to contrast material, pacemakers, claustrophobia, etc.)
25. Have hypersensitivity to dimethyl sulfoxide (DMSO)
26. Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
27. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female patients must undergo a blood or urine pregnancy test at screening and within 36 hours prior to injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment emergent adverse events from the bone marrow-derived allogeneic mesenchymal stem cells implant | At each intervention and 7, 10, and 16 months after last intervention
  Evaluation of treatment emergent adverse events based on viability, safety and tolerance of the bone marrow-derived allogeneic mesenchymal stem cells implant (MSCs) in fistulizing Crohn's Disease patients, defined as:
  * Treatment emergent adverse event (AE) rates, infections, hospitalizations or surgical interventions.
  * Physical examination
  * Vital signs
  * Laboratory tests (biochemistry, hematology, urinalysis)

SECONDARY OUTCOMES:
Clinically: to assess changes in the Crohn's Disease Activity Index (CDAI), the Perianal Disease Activity Index (PDAI). | At each intervention and 7, 10, and 16 months after last intervention
  To monitor the number of draining fistulas, fistula healing efficiency, relapse rate among patients who achieved treatment success and amount local inflammation: Complete closure will be defined as absence of discharge and absence of collections of ≥2 cm directly related to the treated fistulas tracts as assessed by perianal examination. Partial closure will be defined as a reduction in >50% draining fistulas or no discharge on finger compression.
Endoscopic assessment of rectum using a limited simplified endoscopic activity score for Crohn's disease (SES-CD) to evaluate extent and severity of ulcers. | At each intervention and 7, 10, and 16 months after last intervention
  Endoscopic ultrasound and Examination under anesthesia to evaluate baseline fistula state and during each intervention to assess tract closure and abscesses. Remission will be defined as healing of rectal ulcers and/or closure of fistula tracts by endoscopic ultrasonography.
Radiologic assessment using MRI | Baseline, Month 4, and 16 months only if fistula closure has not been achieved at month 4
  to examine number of tracts, inflammation in tracts, and extent of fibrosis or regenerative tissue via MRI assessment. Radiologic remission will be defined as substitution of tracts with fibrosis or regenerative tissue.
Evaluate symptomatic patients. | Month 4 and Month 16
  Endoscopic ultrasound and MRI will be used to evaluate symptomatic patients.
Evaluate the effect of local treatment with allogeneic bmMSCs using the short Inflammatory Bowel Disease Questionnaire (sIBDQ) | At each intervention and 7, 10, and 16 months after last intervention
  To evaluate the effect of local treatment with allogeneic bmMSCs on the quality of life of patients with fistulizing CD using the short Inflammatory Bowel Disease Questionnaire (sIBDQ)
Evaluate the effect of local treatment with allogeneic bmMSCs using the Short Form (SF)-36 score | At each intervention and 7, 10, and 16 months after last intervention
  To evaluate the effect of local treatment with allogeneic bmMSCs on the quality of life of patients with fistulizing CD using the Short Form (SF)-36 score
C-reactive protein (CRP) | At each intervention and 7, 10, and 16 months after last intervention
  To summarize the changes from baseline compared to 12 weeks in serum C-reactive protein
Major Adverse Events | At each intervention and 7, 10, and 16 months after last intervention
  • Incidence of the Major Adverse Events endpoint, defined as the composite incidence of (1) death (2) hospitalization for worsening fistulizing disease (3) or infection caused by the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: David Kerman, MD, Principal Investigator — ISCI / University of Miami

IPD SHARING:
Plan to Share IPD: Undecided